





# IMPROVISATIONAL MUSIC THERAPY (IMT) GUIDELINES

Improvisational music therapy involves the therapist and child spontaneously co-creating music together using singing, playing, and movement. The music therapist follows the child's interests and focus of attention which aims to facilitate the child's social communication development (Geretsegger et al., 2015). Crucially, improvisational music therapy is child-led and aims to facilitate a strong sense of personal agency and autonomy. Previous studies have identified that music engagement is more likely to benefit health and wellbeing when the individual has a greater sense of agency in the musical interaction (Howlin & Rooney, 2021; Howlin, Stapleton & Rooney, 2022; Saarikallio, Randall & Baltazar, 2020; Fritz et al., 2018). However, sessions will also often be carefully structured with improvisations weaving in and out of familiar songs or pre-composed music. During the improvisations, the music therapist may often create a balance between following and leading the child (Oldfield 2006, pp.41-91).

The following guidelines are presented for carrying out IMT sessions with autistic children. It is suggested that these are applied flexibly according to the client within the therapy process. This treatment guide contains information on setting, musical media, goals, and basic principles for treatment.

### Setting

IMT for autistic children is offered in an individual setting. The sessions will occur twice weekly for 30-minute sessions over a 12-week period, in addition to support as usual. The session might need to differ from the chosen duration to meet the needs of the child in the moment if necessary. While some different instruments or activities may be available from session to session, the general physical environment should, if possible, remain consistent and predictable for each individual participant. A core set of instruments will be provided and each therapist may also include others depending on their own preferences and their observations of each child. The music therapist will record the instruments played in each session in the music therapy log. Covers (for example a cloth sheet) will be provided to enable therapists to manage the visual stimulation in busy visual environments. The therapist can drape the sheet over objects that may be distracting for the children.

Each session will be recorded on a video camera provided. The camera must be positioned and set up so that it can capture the sounds and images of both child and music therapist.







#### **Musical Media**

All aspects of musical expression, vocal and instrumental, are used to interact with the child and to assess the child's ability to interact musically and socially. Expression and behaviour that can be perceived in a musical way is also incorporated as a means of interaction in IMT. Precomposed songs or recordings of music may also be used, for example to establish a shared focus of attention, as a starting point for improvised music, or to provide periods of rest in between therapy sequences that may be more demanding for the child due to increased social awareness requirements.

#### Goals

The music therapist will set treatment goals that meet the child's individual needs and specific competences. By choosing individualised developmental goals for each phase of the intervention, the therapist guides the therapy process, enables the child to gradually expand the child's abilities in targeted areas of development, and is also able to evaluate progress and outcomes of therapy. The goals will be recorded in the child's clinical notes, which will be stored onsite, according to each school's policy.

## **Principles**

Listed in the table below is an overview of unique and essential, essential, compatible, and proscribed principles in IMT for children with ASD, and their corresponding rationale, therapist's attitude, activity category, and examples. The table is based both on work done by Geretsegger et al 2015 for the Time A RCT trial and Oldfield's clinical experience in this field (Oldfield 2006, 2016).

| Principle | Purpose/<br>Rationale | Attitude | Category of<br>Activities | Example/<br>Technique |
|---|---|---|---|---|
| Use music making, including improvisation, to provide a holding, reassuring and predictable structure to the sessions. Often | Provide a safe<br>and reassuring<br>environment to<br>enable the child<br>to feel at ease | Tailor and adapt musical offerings to the child's likes and dislikes and mood of the moment. Also make clear endings to a shared activity just before the | Present musical structures with conviction and enthusiasm, while adapting to the needs of the child | A hello song may initially be sung on the guitar but then move to the keyboard to follow the child's interest. A structure may evolve where a gathering drum is |







| | this will involve | | child seems to be | | always played in |
|---|---|---|---|---|---|
| | a "Hello song" or | | losing interest | | one corner of the |
| | greeting activity, | | and needs to | | room, and a |
| | and a prepared | | move on. | | shared |
| | musical ending | | | | improvised piano |
| | | | | | duet is played |
| | | | | | towards the end |
| | | | | | of the session |
| Unique and | | | | | |
| Essential | Engage the child | To motivate the | To use the child's | Think creatively | The therapist may |
| | through | child to attend, | particular musical | about different | bring in an |
| | providing a wide | be present and | interests to widen | ways of using | orchestral |
| | range of musical | interact | the range of | music with each | instrument such |
| | styles, | | musical | child | as the clarinet to |
| | instruments, | | possibilities | | create an |
| | interactions and | | available to the | | improvised |
| | musical games | | therapist and the | | musical exchange |
| | las.ea. gaes | | child | | with the child's |
| | | | Cima | | recorder or reed |
| | | | | | horn playing. |
| | | | To watch, listen | | morni pidymig. |
| | To improvise | To enter into | and be inspired by | To improvise | The therapist may |
| | and engage with | the child's | the child | freely around the | play the keyboard |
| | the child's | world and | the child | child's | to accompany the |
| | movements | provide | | movements, also | child's walking, |
| | movements | motivation for | | incorporating | slowing down and |
| | | the child to | | interactive dance | stopping, to |
| | | interact | | and movement | match the child's |
| | | interact | | exchanges | movements. |
| | | | Follow the child's | excitatiges | movements. |
| | Facilitate | Increase | focus of | Create moments | Dospond to the |
| | Musical and | Increase | | of musical | Respond to the child's utterances |
| | | opportunities | attention, | | |
| | Emotional | for awareness | behaviours, and | attunement/ | and behaviour |
| | Attunement | of self, shared | interests; meet | synchronicity | using improvised |
| | | attention, social | the child where | that may develop | music (e.g., by |
| | | reciprocity, and | they are musically | into emotional | holding, |
| | | relationship | and/or | attunement/ | mirroring, |
| | | building | emotionally | emotional | matching |
| | | | | sharing; | techniques) |
| | | | | incorporate the | |
| | | | | child's interests | |
| | | | | and skills | |

Version 2 23/09/2023







| | Scaffold<br>Interactions<br>Dynamically | Increase<br>opportunities<br>for the child to<br>comprehend,<br>engage in, and<br>initiate<br>interaction | Meet the child's initiatives/ behaviour as communicatively intended | While following the child's lead and musical ideas, form the child's expressions into recognisable musical forms, patterns, or motifs | Apply improvisational music therapy techniques (e.g., rhythmic grounding, shaping, exaggerating, extemporising, frameworking) |
|---|---|---|---|---|---|
| Unique and<br>Essential | Using improvised music making to create a balance between following and initiating | To provide opportunities for interaction, adaptability and negotiation. | To follow the child and enable the child to accept suggestions | The therapist moves in and out of following and initiating to reassure the child but also extend the child's capacity to follow and initiate themselves, and develop interactive skills | The therapist accompanies the child's rhythmic drumming on the keyboard but experiments with slight changes of tempo to encourage joint listening. If the child loses interest or focus the therapist returns to the child's tempo. |
| | Tap into Shared<br>History of<br>(Musical)<br>Interaction | Facilitate<br>predictability/<br>feeling safe and<br>secure | Present as playful<br>and reliable<br>interaction<br>partner fostering<br>the child's range<br>of experience | Affirm the child's expression and actions; jointly create musical/ social motifs and routines | Recognise and repeat the child's expression and actions in an attuned way, giving them a musical form and value |
| | | Facilitate capacity for flexibility/ ability to cope with change | | Create moments<br>where (musical)<br>expectations are<br>playfully violated | Include unexpected pauses and/or dynamic variation in improvised music; redirecting techniques |
| | Provide a Secure<br>Environment | Facilitate predictability/ feeling safe and secure; keep | Present as a reliable and responsible | Provide for consistency in therapy settings | Maintain similar arrangement of objects in therapy room and |

Version 2 23/09/2023







| | | the child's | interaction | | maintain some |
|---|---|---|---|---|---|
| | | anxiety low | partner | | familiarity of instruments |
| | | | | Respond to the child's behaviour in consistent ways | Avoid retreating from interaction partner into "observer" role |
| Essential | | | | Comment on/<br>explain<br>interruptions and<br>unexpected<br>events | If it is necessary<br>to terminate the<br>session, explain<br>why you find it<br>necessary to do<br>so |
| (but not<br>unique to<br>IMT) | Build and<br>Maintain a<br>Positive<br>Therapeutic<br>Relationship | Enable rapport<br>and<br>continuation of<br>therapy | Present with interest, respect, and confidence | Understand/<br>reflect upon<br>meanings of the<br>child's and the<br>therapist's<br>behaviour | Display empathy<br>during (musical)<br>interaction |
| | Follow the<br>Child's Lead<br>(Non-Directive<br>Approach) | Facilitate<br>intrinsic<br>motivation | Follow the child's focus of attention, behaviours, and interests; meet the child where | Incorporate the child's interests and motivations | Relate to a child's<br>preference for<br>numbers in<br>making up a<br>"number song" |
| | | Keep the child's anxiety low | they are musically<br>and/or<br>emotionally | Match level of session/ interaction structure to child's needs | Allow the child to control certain aspects of the interaction; allow the child to functionalise the therapist; offer choices |
| Essential<br>(but not<br>unique to<br>IMT) | Set Treatment<br>Goals | Meet the individual child's needs; guide and evaluate the therapy process | Enable the child<br>to reach the<br>respective next<br>developmental<br>stage in a certain<br>skill area | Assess the child's competences, emerging abilities, and needs; choose intervention strategies and techniques tailored to an | If the child is<br>aware of their<br>own and the<br>therapist's<br>(musical) actions,<br>foster reciprocal<br>interactions |

Version 2 23/09/2023







| | | | | assessed need in a specific area | |
|---|---|---|---|---|---|
| | Facilitate<br>Enjoyment | Increase<br>intrinsic<br>motivation for<br>interaction and<br>opportunities<br>for affect<br>sharing | Present with positive affect, acceptance, affection | Incorporate the child's interests; create pleasant and joyful atmosphere | Display interest in<br>the child and<br>their behaviour<br>and joy during<br>(musical)<br>interaction |
| Compatible<br>(but not<br>necessary) | Adjust Setting According to Families' Needs, Clinical Judgement, and Practical Possibilities | According to generalisation Families' Needs, Clinical everyday Judgement, and Practical support families | Consider the whole range of settings of the child's everyday life | Allow for participation of parents/ caregivers or other family members in the therapy session | Improvise<br>together with the<br>child and a family<br>member in home<br>environment |
| | | | | Employ family<br>member-<br>mediated<br>intervention<br>strategies | Discuss with family members how they can employ musical experiences in interacting with the child; encourage parents to sing and vocalise together with their child |